CLINICAL TRIAL: NCT05746754
Title: Phase II Study of Proton Cranio-spinal Irradiation for Leptomeningeal Metastasis
Brief Title: Proton Cranio-spinal Irradiation for Leptomeningeal Metastasis
Acronym: CSI ProLong
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSI ProLong
Record Dates: First submitted 2023-02-16; First posted 2023-02-28 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-05

CONDITIONS: Leptomeningeal Metastasis
MeSH Terms: conditions — Meningeal Carcinomatosis

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Craniospinal proton radiotherapy (Experimental): 30 Gy in 10 fractions to CNS
  Interventions: Radiation: CSI

INTERVENTIONS:
Radiation: CSI — 30 Gy in 10 fractions to CNS

SUMMARY:
Leptomeningeal metastasis is a rare but serious complication to cancer, with a grave prognosis. No efficient treatment exists.

Recent data suggest that craniospinal radiotherapy lead to superior survival and CNS control compared to focal photon radiotherapy. We want to offer Danish patients the new treatment, but within a protocol, as this is new data with an new treatment principle

DETAILED DESCRIPTION:
Patients must be referred from Danish Departments of Oncology with radiotherapy service.

Patients with leptomeningeal metastasis from both solid and hematological cancers will be offered proton radiotherapy with 30 Gy in 10 fractions to the entire craniospinal axis. Patients will be followed with registration of side effects, neurology and MRI scans every 3 months until 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Metastasis to the leptomeningeal space (LM) surrounding the brain and/ or spinal cord
* Metastasis verified by MRI or CSF cytology
* Karnofsky >=60 (requiring some help, can take care of most personal requirements)
* Adequate bone marrow function

  * Haemoglobin > 5 mmol/l
  * Absolute neutrophil count >1 10^9/l
  * Platelet count > 100 10^9/l
* Patient consent
* Female subjects must either be of non-reproductive potential ( ≥ 60 years old, or with no menses for >1 year without an alternative medical cause], OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a pregnancy test within 2 weeks prior to starting treatment.
* Patient at reproductive potential must agree to practice an effective contraceptive method.

Exclusion Criteria:

* • Previous radiotherapy to the intended treatment site that precludes developing a treatment plan that respects normal tissue tolerances (Yang)

  * Patient with multiple, serious major neurologic deficits per physician/investigator assessment including encephalopathy
  * Patient with extensive systemic disease and without reasonable systemic treatment options
  * Patient who is unable to undergo MRI brain and spine with gadolinium contrast
  * Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
CNS control | 6 months
  local control

SECONDARY OUTCOMES:
overall survival | 1 year
  actuarial
CNS-PFS dependent on tumor site | 1 year
  progression free survival, actuarial
Symptomatology | 1 year
  New symptoms, CTC AE 5.0 grade >=3

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus, Aarhus
  - Department of Oncology, Aalborg University Hospital, Aalborg

IPD SHARING:
Plan to Share IPD: No